CLINICAL TRIAL: NCT04044261
Title: Study of Evoked Emotional Responses for Supporting Research of EMO-001 Device Using Photoplethysmography, Galvanic Skin Response, and Electrocardiography
Brief Title: Study of Evoked Emotional Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monsoon Design Studio LLC (Industry)
Collaborators: Healthark Wellness Solutions LLP (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EMO-001 Phase 0
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Emotion, Expressed
Keywords: Emotional Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Single open-label study arm. All participants are enrolled into this arm.
  Interventions: Procedure: Emotion induction using video

INTERVENTIONS:
Procedure: Emotion induction using video — Emotions are induced in the test subjects using videos in Hindi and English. Each subject is shown three video clips for each of the emotions.

SUMMARY:
Mental health and emotional awareness are a crucial need of the time. Changing lifestyles, stress, and anxiety are seen more commonly and affect many adults in the United States and other countries. Primary aim of this study is to identify the bio-physiological data that is corrected emotions of a person in support of EMO-001 device research.

This study will induce different emotions in the test subjects and collect physiological response signals using Photo Plethysmography (PPG), Galvanic Skin Response (GSR) and Electrocardiogram (ECG) sensors. The sensor data is digitally recorded in a storage bank. The data will be subsequently used to develop supervised and unsupervised classification algorithms.

Emotional states considered in this study are Anger, Amusement, Neutral, Disgust, Sadness, Scared, Surprise and Thrill. These emotions were induced by showing video clips of three to five minutes to the subjects. For each emotion three clips were shown to each subject. Video clips are sourced from movies, TV shows, and real-life recordings. Subjects evaluated each video clip and classify them into perceived emotional ratings.

Data is processed through a series of filter and transformation methods. The transformed data is used to develop and calibrate algorithms that can identify emotions.

DETAILED DESCRIPTION:
Millions of people are affected by mental health conditions every year. Approximately one in five adults in the U.S. experiences at least one mental illness episode every year. Approximately 16 million people have at least one major depressive episode in one year. Researchers have identified that Millennial age-group is at highest risk of developing anxiety, depression, and thoughts of suicide than any other generation. These conditions are attributed by many reasons like increasing competition, less communication, less real-world attachment, work pressure, etc.

Considering the increasing level of issues related to mental health, compelled to think about understanding emotions and associated health impact. Popular methods of emotion detection are by detecting facial expression but to detect real-time emotion, biophysical signals are the best tool as per literature. Also, by considering the future possibility of product form of EMO-001, emotion detection through bio-signals proved to be the correct approach. The intent of the research is to classify the evoked emotions based on bio-signals in support of the product EMO-001 device using photo plethysmography (PPG), Galvanic Skin Response (GSR) and Electrocardiogram (ECG). Identification of emotions from bio-signals, and development of classification algorithm helps the product to identify the emotional state of the person real-time and eventually helps to track the emotional state and suggest an activity which can lift the emotional well being of a person.

Major six emotions, amusement, sad, disgust, scared, surprised, thrill were considered to collect bio signal. Bio signals for the neutral state were also captured to create a baseline for identifying changes in the bio signals with changing emotions.

To find the gender balance in subjects, a similar ratio of male and female considered. Targeting Millennial age-group for this product, we consider people from the age of 18 to 33 years with a minimum bachelor degree qualification and those who are employed. We considered people who understand English and Hindi are considered as subject as video content were in these languages only.

Exploring different methods of emotion elicitation, an audio visual method was considered for this trial, as it is the most effective methods described in different previous literature and through practical scenario. More than 1,000 Video clips from open platform were seen and analysed for five different emotions. Out of which 100 video (20 per emotion) clips were scrutinized by three level checks, selected video clips were also validated by internal blind check to figure out what exact emotion has been elicited from each video. From these identified clips, different set of clips had been prepared. We could identify that video clips are less effective to elicit the anger; hence interaction method was used for it.

Internal validation of data capturing sensors and assembly done to ensure the bio signals obtained are of good quality. For the collection of bio signals, subjects were asked to sit in a proper position, and sensors were placed at particular place of the body.

When the subject was ready for the participation, initially for 30 seconds neutral pictures (e.g. nature sites) were shown to neutralize his/her emotions. After that starting with any of the emotion, three randomly selected videos of a particular emotion from data bank was shown, each followed by a neutral clipping to neutralize the effect of the earlier video. In parallel of videos, the bio-signal data was collected from the sensors. After each video, the subject was asked to fill up a feedback form to rate his emotions. After finishing the signal collection of five different emotions and neutral in between, interaction with subject initiated where the subject was asked about their general background and slowly turned to some sensitive topic which helped to elicit the anger emotion.

The trial had completely non-invasive intervention, where participant need to sit for two hours to watch the videos. Collected data would further be analysed and used for development of emotion classification algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor's degree

Exclusion Criteria:

* History of neurological disorders
* History of psychological disorders
* Current unemployment
* Major surgery in the past two years
* Chronic disease prescriptions

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
ECG V1 | Two hours
  Electrocardiogram V1-lead only
SpO2 | Two hours
  Blood oxygen concentration using photoplethysmography
GSR | Two hours
  Galvanic skin response

CONTACTS AND LOCATIONS:
Overall Officials: Purav Gandhi, MBBS, Principal Investigator — Healthark Wellness Solutions LLP; Anshu Shah, PhD, Study Director — Healthark Wellness Solutions LLP
Locations (1):
- Healthark Wellness Solutions LLP, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No
Data collected is individually identifiable and will not be disclosed to other researchers.